CLINICAL TRIAL: NCT01140789
Title: Genome Wide Association (GWA) Study in Chinese Patients With Inflammatory Bowel Disease
Brief Title: GWA Study in Patients With Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: IBD GWA
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
  1. Up to 50ml of blood sample will be collected and stored at -80°C.
  2. Some blood samples will be sent overseas for DNA extraction and genetic analysis.
     Stool
  3. Stool samples will be collected and stored at -80°C. Some will be analysed with PCR for norovirus and faecal calprotectin in Hong Kong. Some will be sent to Germany for transethnic response mapping.Others will be stored for future analysis.
     Biopsy
  4. For some patients, biopsies from sigmoid will be collected, snap frozen and stored at -80°C, 1 routine biopsy may also be collected for histology. Some will be sent overseas for analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Crohn's disease patients: Diagnosis of Crohn's disease by endoscopy, radiology and histology
- Ulcerative colitis patients: Diagnosis of ulcerative colitis defined by endoscopy, radiology and histology
- Non-IBD patients: Ethically, sex and aged-matched controls attending clinics or endoscopy for functional upper gastrointestinal diseases or screening colonoscopy.

SUMMARY:
The aim of this study is to identify new genes in Chinese patients that help investigators to understand the biological pathway and functions in a population in whom the incidence of Inflammatory Bowel Disease (IBD) is increasing. And to explore the genetic variations in Chinese patients with IBD.

DETAILED DESCRIPTION:
Crohn's disease (CD) and ulcerative colitis (UC) are chronic inflammatory disorders of the gut that cause major life-long disability. Afflicting mostly young people at an age when they are most active both in their private and professional life, inflammatory bowel disease (IBD) represents an important public health problem affecting both the patients education, working abilities, social life . In the past two decades, the incidence and prevalence of CD and UC have been rapidly increasing in Asia. Familial aggregation, twin studies, and recent genetic studies suggest that there is an important genetic component to IBD. In the West, genome wide association (GWA) studies have identified more than 50 genes associated with CD including genes involved in bacterial handling, NOD 2, and the genes involved in autophagy ATG16L1 and IRGM. Only a few of these genes have been studied in Asian populations. Of those which have been studied, such as NOD2, there have been clear differences from Western populations. To date most of the GWA studies have been carried out in cohorts of Caucasian patients. Genetic studies in ethnically different populations may identify new causal variants in IBD, which are likely to lead to further insights into pathophysiology and potential treatments. The aim is to perform a GWA study in Chinese patients with CD and UC. Identifying new genes in Chinese patients will help the investigators to understand the biological pathway and functions in a population in whom the incidence of IBD is increasing. As part of a collaborative project with China, we aim to collect blood samples from 1600 IBD patients and 2000 control subjects in Hong Kong to conduct a GWA study. Samples of 300 IBD patients and 500 controls will be contributed to a collaborative project with China.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Informed consent given by patient or family

Case group (IBD patients) Diagnosis of Crohn's disease or ulcerative colitis defined by endoscopy, radiology and histology

Control group (non-IBD cases) Ethically, sex and aged-matched controls attending clinics or endoscopy for functional upper gastrointestinal diseases or screening colonoscopy.

Exclusion Criteria:

* No consent
* Controls will be excluded if they have previously been diagnosed with IBD or if they have a first or second degree relative with IBD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Crohn's disease or ulcerative colitis patients as the case groups, Patients attend clinics or endoscopy for functional upper gastrointestinal diseases or screening colonoscopy as the control group.
Sampling Method: Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2010-04 (Actual); Primary Completion 2037-04 (Estimated); Study Completion 2037-04 (Estimated)

PRIMARY OUTCOMES:
To identify genetic variation among three study groups | 2 years
  Data will be collected from follow up questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Siew C NG, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No